CLINICAL TRIAL: NCT00343382
Title: Pilocarpine for Vaginal Dryness: A Phase III Randomized, Double Blind, Placebo-Controlled Study
Brief Title: Pilocarpine in Treating Vaginal Dryness in Patients With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N04CA; NCI-2009-00648 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000482969 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Vaginal Dryness
Keywords: sexuality and reproductive issues; sexual dysfunction; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Sexuality; Sexual Dysfunction, Physiological | interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): Patients receive oral pilocarpine hydrochloride once a day for 3 days, twice a day for 3 days, three times a day for 3 days, and then 4 times a day for up to 6 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: pilocarpine hydrochloride
- Arm II (Experimental): Patients receive oral pilocarpine hydrochloride once a day for 3 days and then twice a day for up to 6 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: pilocarpine hydrochloride
- Arm III (Placebo Comparator): Patients receive oral placebo once a day for 3 days, twice a day for 3 days, three times a day for 3 days, and then 4 times a day for up to 6 weeks in the absence of unacceptable toxicity.
  Interventions: Other: placebo
- Arm IV (Placebo Comparator): Patients receive oral placebo once a day for 3 days and then twice a day for up to 6 weeks in the absence of unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: pilocarpine hydrochloride — Given orally
  Arms: Arm I; Arm II
Other: placebo — Given orally
  Arms: Arm III; Arm IV

SUMMARY:
RATIONALE: Pilocarpine may decrease vaginal dryness and improve quality of life in patients with breast cancer It is not yet known whether pilocarpine is more effective than a placebo in treating vaginal dryness in patients with breast cancer.

PURPOSE: This randomized phase III trial is studying pilocarpine to see how well it works compared to a placebo in treating vaginal dryness in patients with breast cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to age (18 to 45 vs 46 to 55 vs 56 to 65 vs > 65), concurrent tamoxifen therapy (yes vs no vs unknown [e.g., on a blinded clinical study]), concurrent aromatase inhibitor therapy (yes vs no vs unknown [e.g., on a blinded clinical study]), and perception of severity of vaginal symptoms at baseline (mild vs moderate vs severe). Patients are randomized to 1 of 4 treatment arms. The primary and secondary objectives of the study are described below.

OBJECTIVES:

Primary

* Determine the effectiveness of pilocarpine hydrochloride for alleviation of vaginal dryness in patients with breast cancer.

Secondary

* Evaluate any toxicities arising from pilocarpine hydrochloride in these patients.
* Evaluate quality of life of these patients treated with pilocarpine hydrochloride.

Quality of life was assessed at baseline and then weekly for 6 weeks.

ELIGIBILITY:
Required Characteristics:

1. Adult post menopausal women or women with no childbearing potential (≥ 18 years) with a history of breast cancer (currently no evidence of disease) or women who do not want to take vaginal estrogen for a fear of an increased risk of breast cancer. Postmenopausal status will be determined by the primary physician.
2. Significant vaginal complaints defined as persistent vaginal dryness and/or itching of sufficient severity to make a patient desire therapeutic intervention. Symptoms should have been present ≥ 2 months prior to randomization.
3. Life expectancy > 6 months
4. Ability to complete questionnaire(s) by themselves or with assistance.

Contraindications:

1. Initiation or discontinuation of tamoxifen or aromatase inhibitors ≤2 months prior to randomization or plans to initiate or discontinue any of these medications during the 6-week study.
2. Active vaginal infection
3. Concurrent chemotherapy
4. Acute iritis
5. Current or past use of pilocarpine (regardless of purpose)
6. Planned use of any vaginal preparations during the study period (including any over the counter or herbal preparations). Note: Lubricants used during sexual intercourse are permitted.
7. Use of any vaginal preparations ≤ 1 week prior to study entry (Exception: If patient has used vaginal preparations during the previous week but will stop, then they can be placed on study with plans to start with pretreatment questionnaire one week later). Note: Lubricants used during sexual intercourse are permitted.
8. Current (≤ 4weeks prior to randomization), or planned during the study period, use of any estrogen product.
9. A diagnosis of asthma, COPD, CAD or narrow angle glaucoma, or known cholelithiasis.
10. Hepatic or renal insufficiency defined as a history of an elevation of SGOT ≥1.5 x ULN or creatinine ≥ 1.5 x ULN within the past year.
11. Concurrent use of other anticholinergics
12. Use of pharmacologic soy preparations
13. Known history of cardiac arrhythmia. (Patients with occasional PVC's or PAC's that do not require treatment are eligible.)
14. Prior or concurrent pelvic radiation therapy
15. Prior radical pelvic surgery (TAH/BSO is allowed)
16. Use of beta adrenergic antagonists
17. Diagnosis of any of the following conditions:

    * Vulvar and vaginal dysplasia
    * Essential vulvodynia
    * Vulvar vestibulitis
    * Vaginal prolapse
    * Bartholin cyst/abscess
    * History of Bartholin gland surgery
    * Lichen sclerosis
    * Lichen planus of the vulvovaginal region
    * Desquamative vaginitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2006-12; Primary Completion 2009-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic
Locations (192):
- United States (192):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin

REFERENCES:
- [Result] Loprinzi CL, Balcueva EP, Liu H, Sloan JA, Kottschade LA, Stella PJ, Carlson MD, Moore DF Jr, Zon RT, Levitt R, Jaslowski AJ. A phase III randomized, double-blind, placebo-controlled study of pilocarpine for vaginal dryness: North Central Cancer Treatment group study N04CA. J Support Oncol. 2011 May-Jun;9(3):105-12. doi: 10.1016/j.suponc.2011.02.005. PMID 21702402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two-hundred and one (201) participants were recruited between December 2006 and May 2009 from 22 North Central Cancer Treatment Group (NCCTG) member sites.
Pre-assignment Details: Five participants (2 collective placebo, 2 Pilocarpine 2 times per day, 1 Pilocarpine 4 times per day) canceled prior to study medication begins and one Pilocarpine 2 times per day participant was ineligible. These six participants were excluded from all analysis.
Groups:
- Collective Placebo: Patients receive 1 capsule of placebo 2 times per day for 6 weeks and; patients receive 1 capsule of placebo 4 times per day for 6 weeks.
- Pilocarpine 2 Times Per Day: Patients receive 5mg of Pilocarpine 2 times per day for 6 weeks.
- Pilocarpine 4 Times Per Day: Patients receive 5mg of Pilocarpine 4 times per day for 6 weeks.
Period: Overall Study
Arm/Group | Collective Placebo | Pilocarpine 2 Times Per Day | Pilocarpine 4 Times Per Day
Started | 64 | 65 | 66
Completed | 60 | 51 | 49
Not Completed | 4 | 14 | 17
Not completed — Adverse Event | 2 | 10 | 7
Not completed — Withdrawal by Subject | 1 | 2 | 6
Not completed — Other Reason Not Specified | 1 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Collective Placebo | Pilocarpine 2 Times Per Day | Pilocarpine 4 Times Per Day | Total
Number analyzed (Participants) | 64 | 65 | 66 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (7.93) | 55.1 (8.14) | 54.7 (7.25) | 54.8 (7.74)
Sex/Gender, Customized [Number; unit: participants]
  Female | 64 | 65 | 66 | 195
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 4
  White | 60 | 63 | 65 | 188
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 64 | 65 | 66 | 195
Tamoxifen use [Number; unit: participants]
  Yes | 10 | 10 | 9 | 29
  No | 54 | 54 | 56 | 164
  Unknown | 0 | 1 | 1 | 2
Current aromatase inhibitor [Number; unit: participants]
  Yes | 36 | 37 | 38 | 111
  No | 28 | 27 | 27 | 82
  Unknown | 0 | 1 | 1 | 2
Severity of vaginal symptoms [Number; unit: participants]
  Mild | 6 | 6 | 6 | 18
  Moderate | 30 | 30 | 30 | 90
  Severe | 28 | 29 | 30 | 87
Breast cancer history [Number; unit: participants]
  Yes | 55 | 59 | 58 | 172
  No | 9 | 6 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Average Vaginal Dryness Scores Via Area Under the Curve (AUC) Summary Statistics
Description: Vaginal dryness was measured by the numerical analogue scale at baseline and through the six weeks of treatment. The item scores was transformed into 0 to 100 scales with 0=poor quality of life (QOL) and 100=best possible QOL. The average AUC values were calculated by dividing 6 from AUC values for participants who completed item on all 6 weeks. If a participant completed the item at baseline, week 1, 2 and 3 but did not complete the item at week 4 to week 6, the AUC values of the item was prorated, which is (((AUC values * 6) / 3) / 6). The average pro-rated AUC for vaginal dryness scores was compared in each of the Pilocarpine arms against the collective placebo arm.
Time Frame: Baseline to Week 6
Population: Includes all participants that reported a baseline value and at least one value after baseline (i.e. week 3, 4, 5 or 6).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collective Placebo | Pilocarpine 2 Times Per Day | Pilocarpine 4 Times Per Day
Number analyzed (Participants) | 61 | 61 | 55
units on a scale | 63.6 (24.04) | 55.8 (27.69) | 66.0 (21.38)
Statistical Analysis 1: Comparison: Collective Placebo vs Pilocarpine 2 Times Per Day; Test type: Superiority or Other; p = 0.1675, Kruskal-Wallis
Statistical Analysis 2: Comparison: Collective Placebo vs Pilocarpine 4 Times Per Day; Test type: Superiority or Other; p = 0.5974, Kruskal-Wallis

2. Secondary Outcome: Toxicity as Measured by Common Terminology Criteria for Adverse Events (CTCAE) 3.0
Description: CTCAE Grading: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening, Grade 5=Death.
Time Frame: End of 6 weeks
Measure: Number; unit: participants
Arm/Group | Collective Placebo | Pilocarpine 2 Times Per Day | Pilocarpine 4 Times Per Day
Number analyzed (Participants) | 63 | 65 | 66
participants
  Grade 1 or 2 rigors | 2 | 14 | 17
  Grade 1 or 2 urinary frequency | 12 | 21 | 29
  Grade 1 or 2 nausea | 7 | 16 | 20
  Grade 1 or 2 sweating | 19 | 29 | 33
Statistical Analysis 1: Comparison: Collective Placebo vs Pilocarpine 2 Times Per Day vs Pilocarpine 4 Times Per Day; Comparison of Rigors among arms; Test type: Superiority or Other; p = 0.002, Kruskal-Wallis
Statistical Analysis 2: Comparison: Collective Placebo vs Pilocarpine 2 Times Per Day vs Pilocarpine 4 Times Per Day; Comparison of Urinary Frequency among arms; Test type: Superiority or Other; p = 0.006, Kruskal-Wallis
Statistical Analysis 3: Comparison: Collective Placebo vs Pilocarpine 2 Times Per Day vs Pilocarpine 4 Times Per Day; Comparison of nausea among arms; Test type: Superiority or Other; p = 0.030, Kruskal-Wallis
Statistical Analysis 4: Comparison: Collective Placebo vs Pilocarpine 2 Times Per Day vs Pilocarpine 4 Times Per Day; Comparison of sweating among arms; Test type: Superiority or Other; p = 0.062, Kruskal-Wallis

3. Secondary Outcome: Average AUC Summary Statistics for the Impact of Vaginal Dryness for Activities of Daily Living
Description: The impact of vaginal dryness for activities of daily living (ADL) were measured by the numerical analogue scales at baseline and through the six weeks of treatment. The item scores was transformed into 0 to 100 scales with 0=poor quality of life (QOL) and 100=best possible QOL. The average AUC values were calculated by dividing 6 from AUC values for participants who completed item on all 6 weeks. If a participant completed the item at baseline, week 1, 2 and 3 but did not complete the item at week 4 to week 6, the AUC values of the item was prorated, which is (((AUC values * 6) / 3) / 6). The average pro-rated AUC scores was compared in each of the Pilocarpine arms against the collective placebo arm.
Time Frame: Baseline to Week 6
Population: Includes all participants that reported a baseline value and at least one value after baseline (i.e. week 3, 4, 5 or 6).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collective Placebo | Pilocarpine 2 Times Per Day | Pilocarpine 4 Times Per Day
Number analyzed (Participants) | 62 | 61 | 55
units on a scale
  Interfered with general activity | 87.9 (15.77) | 87.1 (15.36) | 87.0 (15.72)
  Interfered with mood | 85.4 (17.17) | 75.8 (24.16) | 81.8 (17.65)
  Interfered with normal work | 91.5 (14.08) | 93.0 (11.77) | 92.3 (10.80)
  Interfered with relations with other people | 82.2 (20.62) | 77.9 (25.92) | 80.6 (21.27)
  Interfered with sleep | 93.0 (13.46) | 92.3 (15.81) | 93.3 (9.28)
  Interfered with enjoyment of life | 77.8 (24.24) | 68.7 (27.84) | 76.4 (23.08)

4. Secondary Outcome: Change From Baseline to Week 6 on the Impact of Vaginal Dryness for Activities of Daily Living Scores
Description: The impact of vaginal dryness for activities of daily living (ADL) were measured by the numerical analogue scales at baseline and through the six weeks of treatment. The item scores was transformed into 0 to 100 scales with 0=poor quality of life (QOL) and 100=best possible QOL. The change from baseline scores was calculated by subtracting the baseline item scores from the scores at 6 week.
Time Frame: Baseline and Week 6
Population: Includes all participants who completed both baseline and week 6 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collective Placebo | Pilocarpine 2 Times Per Day | Pilocarpine 4 Times Per Day
Number analyzed (Participants) | 58 | 58 | 54
units on a scale
  Interfered with general activity | 17.8 (26.23) | 16.0 (28.77) | 16.1 (27.02)
  Interfered with mood | 18.3 (29.03) | 17.8 (29.44) | 18.9 (34.62)
  Interfered with normal work | 11.0 (23.15) | 6.0 (18.16) | 9.1 (22.17)
  Interfered with relations with other people | 23.0 (37.41) | 18.5 (33.02) | 24.3 (41.15)
  Interfered with sleep | 5.6 (19.27) | 5.1 (12.75) | 10.8 (21.99)
  Interfered with enjoyment of life | 26.7 (35.17) | 21.1 (36.11) | 30.2 (33.14)

ADVERSE EVENTS:
Time Frame: End of 6 Weeks
Description: Adverse event information at end of 6 weeks is not available on one participant from collective placebo arm.
Arm/Group | Pilocarpine 2 Times Per Day | Pilocarpine 4 Times Per Day | Collective Placebo
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/66 | 0/63
Other Adverse Events (participants affected / at risk) | 48/65 | 47/66 | 33/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilocarpine 2 Times Per Day (N=65) | Pilocarpine 4 Times Per Day (N=66) | Collective Placebo (N=63)
Flashing vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (16) | 20 (20) | 7 (7)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rigors (General disorders) | 14 (14) | 17 (17) | 2 (2)
General symptom (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 10 (10) | 13 (13) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 21 (21) | 29 (29) | 12 (12)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 25 (25) | 14 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 29 (29) | 33 (33) | 19 (19)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes